CLINICAL TRIAL: NCT05889546
Title: Rapid ("Warm") Autopsy Protocol for Patients With Small Cell Lung Cancer
Brief Title: Rapid Autopsy Protocol for Patients With Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shadia Jalal, Associate Professor in the Department of Medicine at Indiana University, Indiana University
Other Study IDs: CTO-IUSCCC-0783
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Lung Cancer; Small Cell Lung Cancer; Future Research
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active SCLC Diagnosis
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Lung, liver, skin, subcutaneous metastases, and blood specimens may be collected via rapid autopsy within 10 hours of expiration.

SUMMARY:
This is pilot study to establish a rapid autopsy program in Small Cell Lung Cancer (SCLC) at the Indiana University Simon Comprehensive Cancer Center and outline the components necessary for tumor tissue collection.

DETAILED DESCRIPTION:
The goal of this project to establish a rapid autopsy program in SCLC at the IUSCCC and outline the key components necessary for tumor tissue acquisition. This proposal is a collaboration between scientists, lung cancer physicians, pathologists, and the IUSCCC Translational Research Core. Tumor tissue collected will be used for protein and gene analysis and RNA, whole exome sequencing in addition to the establishment of SCLC. This research is part of a discovery project in which biological and molecular markers of SCLC will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Written informed consent and HIPAA authorization for release of personal health information.
3. Active SCLC diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with active SCLC being seen at IUSCCC clinics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining the Feasibility of the Creation of a Rapid Autopsy Program at IUSCCC for SCLC through enrollment and sample collections | 5 years
Utilization of Tissue to Better Understand the Complex Biology of SCLC | 5 years
  Utilize tissue obtained from rapid autopsies to generate novel patient derived xenograft models and tumor cell lines, in addition to RNA, whole exome and whole genome sequencing, protein extraction to better understand the complex biology of SCLC and set up an infrastructure to develop relevant clinical models that will allow the development of better therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia I. Jalal, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Roudebush VA Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana